CLINICAL TRIAL: NCT00551187
Title: A Randomized, Double-Blinded, Tolerability and Immunogenicity Study of a Multivalent Human Papillomavirus (HPV) L1 Virus-Like Particle (VLP) Vaccine Administered Concomitantly With GARDASIL to 16- to 26- Year-Old Women
Brief Title: A Study to Evaluate Tolerability and Immunogenicity of V504 Administered Concomitantly With GARDASIL (V504-001)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V504-001; 2007_566
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Cervical Cancer; Vulvar Cancer; Vaginal Cancer; Genital Warts; Human Papillomavirus Infection
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Condylomata Acuminata; Papillomavirus Infections | interventions — Vaccines, Synthetic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): V504 + Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine
  Interventions: Biological: V504; Biological: Comparator: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine
- 2 (Placebo Comparator): Placebo + Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine
  Interventions: Biological: Comparator: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine; Biological: Comparator: Placebo (unspecified)

INTERVENTIONS:
Biological: V504 — V504 0.5 ml injection in 3 dose regimen for 6 month treatment period.
  Arms: 1
Biological: Comparator: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine — Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine 0.5 ml injection in 3 dose regimen for 6 month treatment period.
Biological: Comparator: Placebo (unspecified) — V504 Placebo in 3 dose regimen for 6 month treatment period.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate vaccine immunogenicity and how well the body tolerates V504 when given with Gardasil.

ELIGIBILITY:
Inclusion Criteria:

* Females between 16- to 26-years-old
* Has never had Pap testing or has only had normal Pap test results.
* Lifetime history of 0 to 4 sexual partners

Exclusion Criteria:

* History of an abnormal cervical biopsy result
* History of a positive test for HPV; History of external genital/vaginal warts
* Currently a user of illegal drugs or an alcohol abuser
* History of severe allergic reaction that required medical attention
* Are pregnant
* Received a marketed HPV vaccine
* Currently enrolled in a clinical trial
* Currently has or has a history of certain medical conditions or is currently taking or has taken certain medications (details will be discussed at the time of consent)

Ages: 16 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 620 (Actual)
Dates: Start 2007-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Geometric mean titers (GMTs) to HPV types contained in the administered vaccines | 4 weeks post dose 3

SECONDARY OUTCOMES:
Seroconversion percentages to HPV types contained in the administered vaccines | 4 weeks post dose 3

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Luxembourg A, Brown D, Bouchard C, Giuliano AR, Iversen OE, Joura EA, Penny ME, Restrepo JA, Romaguera J, Maansson R, Moeller E, Ritter M, Chen J. Phase II studies to select the formulation of a multivalent HPV L1 virus-like particle (VLP) vaccine. Hum Vaccin Immunother. 2015;11(6):1313-22. doi: 10.1080/21645515.2015.1012010. PMID 25912208